CLINICAL TRIAL: NCT04783051
Title: Comparison of IST Using Ultra-sensitive Malaria Rapid Diagnostic Test and Pyronaridine - Artesunate - PYRAMAX®) to Standard IPT Sulfadoxine-pyrimethamine to Prevent Malaria in Pregnant Women Living in Endemic Areas
Brief Title: Comparison of ISTp- PYRAMAX-US-RDT to IPTp-SP to Prevent Malaria in Pregnant Women in DRC (ULTRAPYRAPREG)
Acronym: ULTRAPYRAPREG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kinshasa (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Novartis (Industry)
Responsible Party: Principal Investigator, Vivi Maketa, Professor, University of Kinshasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 226/CNES/BN//PMMF/2020
Record Dates: First submitted 2021-02-27; First posted 2021-03-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Malaria in Pregnancy
Keywords: Malaria; Pregnancy; IPTp-SP; ISTp-Pyramax; Kinshasa; DR Congo
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPTp-SP (Active Comparator): The IPTp-SP group will be pregnant women who will receive the standard regimen recommended by the Malaria National Control Program (MNCP) at week 16, 28, 32 and 36 of their pregnancy
  Interventions: Drug: Sulfadoxine pyrimethamine
- ISTp-US-Py (Experimental): The ISTp-US-Py group will comprise pregnant women who will be screened monthly from the beginning of the 2nd trimester with ultra-sensitive -RDT and who will be treated with Pyramax® if the test is positive
  Interventions: Drug: Pyramax

INTERVENTIONS:
Drug: Sulfadoxine pyrimethamine — Intermittent Preventive Treatment in pregnant women with Sulfadoxine-Pyrimethamine
  Other Names: IPTp-SP
  Arms: IPTp-SP
Drug: Pyramax — Intermittent screening using ultra-sensitive malaria Rapid Diagnostic test and treatment using Pyronaridine - Artesunate (PYRAMAX®)
  Other Names: ISTp-US-Py
  Arms: ISTp-US-Py

SUMMARY:
In endemic settings Plasmodium falciparum (Pf) can sequester in the placenta resulting in low peripheral parasitemia and false negative malaria diagnosis in pregnant women. Intermittent Preventive Treatment in pregnant women with Sulphadoxine-Pyrimethamine (IPTp-SP) is one of the World Health Organization's recommended malaria control strategies in sub-Saharan African countries. The strategy overcomes the risk of misdiagnosis of malaria in pregnant women by treating them all with SP according to predetermined schedules, but the strategy is now threatened by the spread of Plasmodium parasite resistant strains. As a necessary alternative, Intermittent Screening and Treatment in pregnancy (ISTp), aims on the monthly screening of pregnant women with a malaria rapid diagnostic test (RDT) and the treatment of positive cases with artemisinin-based combination therapy (ACT) regardless of the presence of symptoms. The ISTp depends on the performance of the diagnostic tests, and the use of ultrasensitive RDTs (us-RDTs), which have a higher analytical sensitivity than conventional RDTs, should improve the efficacy of the strategy.

Unlike IPTp-SP, ISTp prevents overuse of antimalarials and thus limits drug pressure on malaria parasites. This advantage could be potentiated by using, for pregnant women, an ACT that is not yet used or should not be used in the field for other strata of the population. The recently approved new ACT combination, Pyronaridine - Artesunate (Pyramax®) is the ideal candidate for this purpose.

This study will compare the effects of the ISTp using an us-RDT and Pyramax® (ISTp-US-Py) with the standard IPTp-SP on maternal malaria indicators (malaria infection, parasite density), maternal anemia, spontaneous abortions or intrauterine deaths during pregnancy, fetal morbidity (preterm birth, low birth weight, small for gestational age) and neonatal mortality at delivery in both study groups through conducting a randomized clinical trial enrolling second trimester pregnant women in Maternité Esengo Health Center, located in Kisenso, Kinshasa, the Democratic Republic of the Congo (DRC), a malaria perennial transmission area.

The results generated from this study will be essential for the National Malaria Control Program in the selection and implementation of new malaria control policies and addresses the effectiveness of IPTp-SP decline among pregnant women in the DRC.

DETAILED DESCRIPTION:
1. Introduction Malaria is a threat for pregnant women and their offspring in endemic settings (1, 2). Plasmodium falciparum (Pf) can sequester in the placenta during pregnancy, resulting in low peripheral parasitemia. As a consequence, malaria diagnostic tests are often false negative in pregnant women who actually do have a Pf malaria infection (3, 4).

Intermittent Preventive Treatment in pregnant women with Sulfadoxine-Pyrimethamine (IPTp-SP) is one of the World Health Organization (WHO)'s recommended malaria control strategies in sub-Saharan African countries (2). The IPTp-SP strategy surmounts the potential misdiagnosis of malaria in pregnant women by treating them all with SP at pre-determined schedules during the antenatal care (ANC) visits. The efficacy of IPTp-SP is dose dependent and relies on ANC coverage. However, the spread of Plasmodium SP resistant strains now threatens the efficacy of the IPTp-SP and can lead to the proliferation of placental resistant parasites in pregnant women (5-9).

As an alternative for IPTp-SP, Intermittent Screening and Treatment in pregnancy (ISTp) may be considered as an option (10). ISTp comprises of monthly screening of pregnant women with a malaria RDT and treatment of positive cases with an artemisinin-based combination therapy (ACT) regardless of the presence of symptoms. The ISTp depends on the performance of the diagnostic tests and the use of ultrasensitive RDTs (us-RDTs), which have a higher sensitivity than conventional RDTs (11, 12), can avoid false negative that would prevent the method from being effective.

Unlike IPTp-SP, ISTp prevents overuse of antimalarials and, thus, limits drug pressure on malaria parasites (10). This advantage could be potentiated by using an ACT that is not yet used or should not be used by the national malaria control for other strata of the population than pregnant women. Pyronaridine - Artesunate (Pyramax®), a newly approved antimalarial is the ideal candidate for this purpose in Democratic Republic of Congo (DRC). Pyramax®, approved for use in malaria endemic countries since 2015, is used in the field to treat malaria in children and adults (13). There is little information on the safety of Pyramax® during pregnancy, however, Pyronaridine unintentionally administered successfully treated at least 40 cases of malaria in late pregnancy (14) and, a review reported that ACTs, although Pyramax® was not included in, are generally very effective and well tolerated during the second and third trimesters (15).

The hypothesis of this study is that the ISTp using Pyramax® for the treatment and performed with the us-RDT (ISTp-US-Py) is non inferior than IPTp-SP for the prevention of maternal malaria (malaria infection, parasite density), maternal anemia, spontaneous abortions or intrauterine death during pregnancy, fetal morbidity (premature birth, low birth weight, small for gestational age) and neonatal mortality at childbirth.

ELIGIBILITY:
Inclusion Criteria:

1. Gestation ≥16 weeks;
2. Age: ≥18 years;
3. Residence within the health facility catchment area;
4. Willing to adhere to study requirements and to deliver at the health facility.
5. Willing to provide written informed consent; if the woman is illiterate, she can choose an impartial witness, not related to the study, to accompany her during the informant consent process and they will both sign the informed consent form

Exclusion Criteria:

1. Known history of allergy to SP or to an ACT
2. An ongoing antibioprophylaxis with cotrimoxazole,
3. Current issue requiring hospital admission (including severe malaria as defined by WHO)
4. Pregnancy at high risk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 250 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
The proportion of asymptomatic malaria in the 2 study arms | 6 months
  Asymptomatic malaria is defined as the presence of Pf diagnosed by an us-RDT in the peripheral blood and a T°≤38°C
The proportion symptomatic malaria in the 2 study arms | 6 months
  Symptomatic malaria is be defined as the presence of Pf diagnosed by an us-RDT in the peripheral blood and a T°≥38°C
The proportion of parasitic densities in the 2 study arms | 6 months
  Parasite density is assessed by the quantification of Pf parasites in the peripheral blood of asymptomatic/symptomatic women by a thin blood smear examined by standard malaria microscopy
The proportion of anemia in the 2 study arms | 6 months
  Anemia is defined as a level of hemoglobin (Hb) <10g/dl
The incidence of spontaneous abortions or intrauterine deaths in the 2 study arms | 6 months
  Intrauterine death is defined to describe the death of the offspring in the uterus
The proportion of fetal morbidities in the 2 study arms | 6 months
  Fetal morbidity is defined as any of the following: Preterm birth (birth before 37 weeks gestation) and low-birth-weight (birth weight under 2,500 grams)
The proportion of the neonatal and early neonatal mortality of the offspring in the 2 study arms | 28 days
  The early neonatal mortality is defined as infant death at birth or within 7 days of life; And the neonatal mortality is defined as infant death within the first 28 days of life

CONTACTS AND LOCATIONS:
Locations (1):
- Maternité Esengo, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Document to be share: all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting right after the publication
Access Criteria: Data will be shared with any researcher who will ask via any contact of the corresponding author of any publication resulting from this clinical trial

REFERENCES:
- [Background] Nosten F, McGready R, Mutabingwa T. Case management of malaria in pregnancy. Lancet Infect Dis. 2007 Feb;7(2):118-25. doi: 10.1016/S1473-3099(07)70023-3. PMID 17251082
- [Background] WHO. Guidelines for the treatment of malaria. Third edition2015. 316 p
- [Background] Anchang-Kimbi JK, Achidi EA, Nkegoum B, Sverremark-Ekstrom E, Troye-Blomberg M. Diagnostic comparison of malaria infection in peripheral blood, placental blood and placental biopsies in Cameroonian parturient women. Malar J. 2009 Jun 8;8:126. doi: 10.1186/1475-2875-8-126. PMID 19505312
- [Background] Matangila JR, Lufuluabo J, Ibalanky AL, Inocencio da Luz RA, Lutumba P, Van Geertruyden JP. Asymptomatic Plasmodium falciparum infection is associated with anaemia in pregnancy and can be more cost-effectively detected by rapid diagnostic test than by microscopy in Kinshasa, Democratic Republic of the Congo. Malar J. 2014 Apr 2;13:132. doi: 10.1186/1475-2875-13-132. PMID 24690179
- [Background] van Eijk AM, Hill J, Larsen DA, Webster J, Steketee RW, Eisele TP, ter Kuile FO. Coverage of intermittent preventive treatment and insecticide-treated nets for the control of malaria during pregnancy in sub-Saharan Africa: a synthesis and meta-analysis of national survey data, 2009-11. Lancet Infect Dis. 2013 Dec;13(12):1029-42. doi: 10.1016/S1473-3099(13)70199-3. Epub 2013 Sep 18. PMID 24054085
- [Background] WHO. World Malaria Report 2017. Geneva: World Health Organization; 2017
- [Background] Harrington WE, Mutabingwa TK, Kabyemela E, Fried M, Duffy PE. Intermittent treatment to prevent pregnancy malaria does not confer benefit in an area of widespread drug resistance. Clin Infect Dis. 2011 Aug 1;53(3):224-30. doi: 10.1093/cid/cir376. PMID 21765070
- [Background] McGready R, White NJ, Nosten F. Parasitological efficacy of antimalarials in the treatment and prevention of falciparum malaria in pregnancy 1998 to 2009: a systematic review. BJOG. 2011 Jan;118(2):123-35. doi: 10.1111/j.1471-0528.2010.02810.x. PMID 21159117
- [Background] Cottrell G, Moussiliou A, Luty AJ, Cot M, Fievet N, Massougbodji A, Deloron P, Tuikue Ndam N. Submicroscopic Plasmodium falciparum Infections Are Associated With Maternal Anemia, Premature Births, and Low Birth Weight. Clin Infect Dis. 2015 May 15;60(10):1481-8. doi: 10.1093/cid/civ122. Epub 2015 Feb 18. PMID 25694651
- [Background] Esu E, Berens-Riha N, Pritsch M, Nwachuku N, Loescher T, Meremikwu M. Intermittent screening and treatment with artemether-lumefantrine versus intermittent preventive treatment with sulfadoxine-pyrimethamine for malaria in pregnancy: a facility-based, open-label, non-inferiority trial in Nigeria. Malar J. 2018 Jul 6;17(1):251. doi: 10.1186/s12936-018-2394-2. PMID 29976228
- [Background] Das S, Jang IK, Barney B, Peck R, Rek JC, Arinaitwe E, Adrama H, Murphy M, Imwong M, Ling CL, Proux S, Haohankhunnatham W, Rist M, Seilie AM, Hanron A, Daza G, Chang M, Nakamura T, Kalnoky M, Labarre P, Murphy SC, McCarthy JS, Nosten F, Greenhouse B, Allauzen S, Domingo GJ. Performance of a High-Sensitivity Rapid Diagnostic Test for Plasmodium falciparum Malaria in Asymptomatic Individuals from Uganda and Myanmar and Naive Human Challenge Infections. Am J Trop Med Hyg. 2017 Nov;97(5):1540-1550. doi: 10.4269/ajtmh.17-0245. Epub 2017 Aug 18. PMID 28820709
- [Background] Vasquez AM, Medina AC, Tobon-Castano A, Posada M, Velez GJ, Campillo A, Gonzalez IJ, Ding X. Performance of a highly sensitive rapid diagnostic test (HS-RDT) for detecting malaria in peripheral and placental blood samples from pregnant women in Colombia. PLoS One. 2018 Aug 2;13(8):e0201769. doi: 10.1371/journal.pone.0201769. eCollection 2018. PMID 30071004
- [Background] Ayyoub A, Methaneethorn J, Ramharter M, Djimde AA, Tekete M, Duparc S, Borghini-Fuhrer I, Shin JS, Fleckenstein L. Population Pharmacokinetics of Pyronaridine in Pediatric Malaria Patients. Antimicrob Agents Chemother. 2015 Dec 14;60(3):1450-8. doi: 10.1128/AAC.02004-15. PMID 26666916
- [Background] Croft SL, Duparc S, Arbe-Barnes SJ, Craft JC, Shin CS, Fleckenstein L, Borghini-Fuhrer I, Rim HJ. Review of pyronaridine anti-malarial properties and product characteristics. Malar J. 2012 Aug 9;11:270. doi: 10.1186/1475-2875-11-270. PMID 22877082
- [Background] D'Alessandro U, Hill J, Tarning J, Pell C, Webster J, Gutman J, Sevene E. Treatment of uncomplicated and severe malaria during pregnancy. Lancet Infect Dis. 2018 Apr;18(4):e133-e146. doi: 10.1016/S1473-3099(18)30065-3. Epub 2018 Jan 31. PMID 29395998
- [Background] West African Network for Clinical Trials of Antimalarial Drugs (WANECAM). Pyronaridine-artesunate or dihydroartemisinin-piperaquine versus current first-line therapies for repeated treatment of uncomplicated malaria: a randomised, multicentre, open-label, longitudinal, controlled, phase 3b/4 trial. Lancet. 2018 Apr 7;391(10128):1378-1390. doi: 10.1016/S0140-6736(18)30291-5. Epub 2018 Mar 29. PMID 29606364
- [Derived] Tshiongo JK, Khote FL, Kabena M, Mavoko HM, Kalonji-Mukendi T, Luzolo L, Schallig HDFH, Kayentao K, Mens PF, Lutumba P, Tinto H, Maketa V. Intermittent screening using ultra-sensitive malaria rapid diagnostic test and treatment with pyronaridine-artesunate compared to standard preventive treatment with sulfadoxine-pyrimethamine for malaria prevention in pregnant women in Kinshasa, DRC. Malar J. 2025 Feb 21;24(1):58. doi: 10.1186/s12936-025-05260-6. PMID 39985024
- [Derived] Maketa V, Kabalu J, Kabena M, Luzolo F, Muhindo-Mavoko H, Schallig HDFH, Kayentao K, Mens PF, Lutumba P, Tinto H. Comparison of intermittent screening (using ultra-sensitive malaria rapid diagnostic test) and treatment (using a newly registered antimalarial pyronaridine-artesunate-PYRAMAX(R)) to standard intermittent preventive treatment with sulfadoxine-pyrimethamine for the prevention of malaria in pregnant women living in endemic areas: ULTRAPYRAPREG. Trials. 2022 Nov 28;23(1):963. doi: 10.1186/s13063-022-06884-8. PMID 36443882
- See also: The PYRAPREG project — https://www.pyrapreg.org/about-project/
- See also: Clinical trials and operational research studies to optimise the use of products for poverty-related diseases in mothers, newborns, children and/or adolescents — https://www.era-learn.eu/network-information/networks/edctp-ii/clinical-trials-and-operational-research-studies-to-optimise-the-use-of-products-for-poverty-related-diseases-in-mothers-newborns-children-and-or-adolescents/efficacy-and-safety-of-a-newly-registered-artemisinin-based-combination-pyronaridine-artesunate-pyramax-r-for-the-treatment-of-uncomplicated-malaria-in-african-pregnant-women
- See also: Pharmaceuticals R. FANSIDAR. brand of sulfadoxine and pyrimethamine TABLETS 1996 — https://www.accessdata.fda.gov/drugsatfda_docs/label/2004/18557slr015_fansidar_lbl.pdf